CLINICAL TRIAL: NCT07152145
Title: Transcutaneous Electrical Spinal Stimulation (tSCS) for Improving Upper Limb Function in People With MS
Brief Title: Pilot Study of tSCS for Improving Upper Limb Function in People With Multiple Sclerosis
Acronym: tSCS-MS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, PAblo Villoslada, Principal Investigator, Neurology Department, Hospital del Mar Research Institute, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: tSCS-MS-01
Record Dates: First submitted 2025-08-22; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Multiple Sclerosis
Keywords: Spinal Cord Neuromodulation; Non-invasive neuromodulation; Upper limb function; Neurorehabilitation
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Active tSCS + Rehabilitation (Experimental): Participants will receive active transcutaneous spinal cord stimulation (tSCS) using the SCONE™ device, combined with conventional upper limb rehabilitation therapy.
  Interventions: Device: Active stimulation tSCS; Behavioral: Occupational/Upper Limb Rehabilitation Therapy
- Sham tSCS + Rehabilitation (Sham Comparator): Participants will receive sham stimulation using the SCONE™ device without active current, combined with conventional upper limb rehabilitation therapy. The setup will be identical to the active intervention to maintain blinding.
  Interventions: Device: Sham: stimulations using a non-active electric stimulation; Behavioral: Occupational/Upper Limb Rehabilitation Therapy

INTERVENTIONS:
Device: Active stimulation tSCS — Active transcutaneous spinal cord stimulation (tSCS) delivered with the SCONE™ device. Electrical currents are applied non-invasively through surface electrodes placed on the skin over the spine. Sessions are combined with standardized upper limb rehabilitation therapy. Participants receive stimulation twice per week for 12 weeks.
  Arms: Active tSCS + Rehabilitation
Device: Sham: stimulations using a non-active electric stimulation — Sham stimulation delivered with the SCONE™ device, using identical setup and procedures as the active intervention but without effective current. This procedure is designed to mimic the sensation and experience of active stimulation while delivering no therapeutic neuromodulation. Participants also perform standardized upper limb rehabilitation therapy twice per week for 12 weeks.Transcutaneous Spinal Cord Stimulation (tSCS) - Sham (SCONE™)
  Arms: Sham tSCS + Rehabilitation
Behavioral: Occupational/Upper Limb Rehabilitation Therapy — Standardized occupational therapy program focused on upper limb function. Sessions are delivered in combination with either active or sham transcutaneous spinal cord stimulation.

SUMMARY:
The goal of this clinical trial is to evaluate whether non-invasive spinal cord neuromodulation with the SCONE™ device can improve upper limb function in people with multiple sclerosis. The study will investigate if combining SCONE™ therapy with rehabilitation exercises leads to improvements in arm and hand movement, and whether the therapy is safe and well tolerated in this patient population. Participants will receive non-invasive spinal cord stimulation with the SCONE™ device and perform rehabilitation exercises specifically focused on the upper limb.

DETAILED DESCRIPTION:
This is a pilot, randomized, placebo-controlled study designed to evaluate the efficacy and safety of transcutaneous spinal cord stimulation (tSCS) in improving upper limb function in patients with Multiple Sclerosis (MS).

tSCS is a non-invasive neuromodulation technique that delivers low-intensity electrical impulses through the skin to specific spinal segments. This external stimulation aims to enhance spinal excitability and restore communication between the brain and spinal circuits affected by MS. Previous research in spinal cord injury has demonstrated functional improvements in motor performance with tSCS, suggesting its potential benefit in MS-related disability.

In this study, participants with clinically confirmed MS and upper limb impairment will first undergo a 6-week period of standard occupational therapy. After this run-in phase, they will be randomly assigned in a 1:1 ratio to receive either active tSCS or sham stimulation for an additional 6 weeks, while continuing occupational therapy. The intervention will be delivered at the rehabilitation center of Hospital de la Esperanza, in a seated position, using surface electrodes placed at the posterior cervical region. Sessions will last approximately 30 minutes, three times per week (preferably Monday, Wednesday, and Friday).

The sham condition will mimic the procedure using the same equipment and electrode placement but without delivering effective stimulation. After completion of the blinded phase, participants originally randomized to sham will be offered the opportunity to receive active tSCS in an open-label extension.

The primary efficacy endpoint is improvement in upper limb function, assessed by the Nine-Hole Peg Test (9HPT). Secondary endpoints include the Action Research Arm Test (ARAT), patient-reported outcomes (NeuroQOL - Upper Extremity Function, Modified Fatigue Impact Scale [MFIS], and Global Impression of Change [GIC]), and clinical safety measures.

tSCS is generally safe and well-tolerated. Reported side effects are typically mild and transient, including tingling, skin irritation, or muscle discomfort. Participants will be monitored throughout the study, and adverse events will be recorded.

This pilot trial will provide preliminary data on the clinical utility of tSCS in MS and inform the design of larger randomized controlled trials.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years.
* Diagnosis of Multiple Sclerosis (according to revised McDonald criteria).
* Upper limb dysfunction (9-Hole Peg Test score ≥ 20% slower than normative values).
* Stable disease-modifying treatment for ≥ 6 months before enrollment.
* Expanded Disability Status Scale (EDSS) score between 3.0 and 6.5.
* Ability to provide informed consent.

Exclusion Criteria:

* Relapse or corticosteroid treatment within the last 3 months.
* Severe spasticity of the upper limb (Modified Ashworth Scale > 3).
* Implanted electrical devices (pacemaker, spinal cord stimulator).
* Epilepsy or uncontrolled seizures.
* Severe psychiatric disorders or cognitive impairment interfering with study procedures.
* Pregnant or breastfeeding women.
* Participation in another interventional clinical trial within the last 3 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Upper Limb Function (9-Hole Peg Test) | Baseline and Week 12
  The 9-Hole Peg Test (9HPT) is a validated quantitative measure of upper extremity function. Participants are timed while placing and removing nine pegs into holes on a board as quickly as possible. Performance is recorded as time to completion. Change from baseline will be compared between active and sham groups.

SECONDARY OUTCOMES:
Change in Hand Grip Strength (Dynamometry) | Baseline and Week 12
  Grip strength will be measured using a calibrated hand dynamometer. The mean of three trials per hand will be recorded and analyzed as change from baseline.
Change in Quality of Life (EQ-5D-5L) | Baseline and Week 12
  Patient-reported outcome measuring five domains of health-related quality of life (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Change from baseline will be assessed.
Change in Fatigue (Modified Fatigue Impact Scale - MFIS) | Baseline and Week 12
  Self-reported questionnaire measuring the impact of fatigue on physical, cognitive, and psychosocial functioning. Change from baseline will be analyzed.
Change in Manual Dexterity (Box and Block Test) | Baseline and Week 12
  The Box and Block Test measures gross manual dexterity by counting the number of blocks moved from one compartment to another in 60 seconds. Change from baseline will be assessed
Patient-Reported Upper Limb Function (Multiple Sclerosis Impact Scale - MSIS-29, upper limb subitems) | Baseline and Week 12
  Patient-reported outcome measure assessing the perceived impact of MS on physical function, with specific focus on upper limb-related items. Higher scores indicate greater impact. Change from baseline will be compared.
Safety and Tolerability | Baseline through Week 12
  Number and severity of adverse events related to the device or therapy will be recorded throughout the study. Tolerability will be assessed via patient-reported discomfort during stimulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital del Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in future publications will be shared. This will include baseline characteristics, efficacy outcomes, and safety data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: IPD and supporting documents will be available within 12 months after publication of the main results and will remain available for a minimum of 5 years thereafter.
Access Criteria: Access will be granted to qualified researchers with a sound scientific proposal for secondary analyses related to multiple sclerosis or neuromodulation. Requests will be reviewed by the study steering committee. Data will be shared through a secure data-sharing platform after signing a data access agreement to ensure confidentiality and appropriate use.

REFERENCES:
- [Background] Inanici F, Samejima S, Gad P, Edgerton VR, Hofstetter CP, Moritz CT. Transcutaneous Electrical Spinal Stimulation Promotes Long-Term Recovery of Upper Extremity Function in Chronic Tetraplegia. IEEE Trans Neural Syst Rehabil Eng. 2018 Jun;26(6):1272-1278. doi: 10.1109/TNSRE.2018.2834339. PMID 29877852
- [Background] Moritz C, Field-Fote EC, Tefertiller C, van Nes I, Trumbower R, Kalsi-Ryan S, Purcell M, Janssen TWJ, Krassioukov A, Morse LR, Zhao KD, Guest J, Marino RJ, Murray LM, Wecht JM, Rieger M, Pradarelli J, Turner A, D'Amico J, Squair JW, Courtine G. Non-invasive spinal cord electrical stimulation for arm and hand function in chronic tetraplegia: a safety and efficacy trial. Nat Med. 2024 May;30(5):1276-1283. doi: 10.1038/s41591-024-02940-9. Epub 2024 May 20. PMID 38769431
- [Background] Tu YH, Stiles ML, Allen LV Jr, Olsen KM, Barton CI, Greenwood RB. Stability of amoxicillin trihydrate-potassium clavulanate in original containers and unit dose oral syringes. Am J Hosp Pharm. 1988 May;45(5):1092-9. PMID 3400652
- [Background] Barss TS, Parhizi B, Porter J, Mushahwar VK. Neural Substrates of Transcutaneous Spinal Cord Stimulation: Neuromodulation across Multiple Segments of the Spinal Cord. J Clin Med. 2022 Jan 27;11(3):639. doi: 10.3390/jcm11030639. PMID 35160091
- [Background] Waltz JM, Andreesen WH, Hunt DP. Spinal cord stimulation and motor disorders. Pacing Clin Electrophysiol. 1987 Jan;10(1 Pt 2):180-204. doi: 10.1111/j.1540-8159.1987.tb05947.x. PMID 2436177
- [Background] Wallin MT, Culpepper WJ, Campbell JD, Nelson LM, Langer-Gould A, Marrie RA, Cutter GR, Kaye WE, Wagner L, Tremlett H, Buka SL, Dilokthornsakul P, Topol B, Chen LH, LaRocca NG; US Multiple Sclerosis Prevalence Workgroup. The prevalence of MS in the United States: A population-based estimate using health claims data. Neurology. 2019 Mar 5;92(10):e1029-e1040. doi: 10.1212/WNL.0000000000007035. Epub 2019 Feb 15. PMID 30770430

DOCUMENTS (2):
  • Study Protocol (2025-05-11): https://cdn.clinicaltrials.gov/large-docs/45/NCT07152145/Prot_000.pdf
  • Informed Consent Form (2025-04-14): https://cdn.clinicaltrials.gov/large-docs/45/NCT07152145/ICF_001.pdf